CLINICAL TRIAL: NCT03806023
Title: EMG Triggered Closed-Loop Stimulation for Spinal Cord Injury Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding expired due to grant for new project (NCT03851302)
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Noam Y. Harel, Principal Investigator, Bronx VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Wu-17-18
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injuries
Keywords: transcutaneous electric nerve stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All subjects (Experimental): All subjects undergo same full protocol, including PNS and TMS at rest and active hand movements (signals from thumb muscle) triggered PNS and TMS.
  Interventions: Device: hand movements (signals from thumb muscle) triggered PNS and TMS

INTERVENTIONS:
Device: hand movements (signals from thumb muscle) triggered PNS and TMS — PNS, TMS or PNS+TMS will be delivered while the participant performs specific finger tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.

SUMMARY:
Most individuals with spinal cord injury (SCI) have residual nerve circuits. The investigators aim to strengthen those circuits to improve motor recovery after injury. To do this, the investigators are attempting to pair electrical and magnetic stimulation with physical training targeted toward the connections between nerve circuits. Past studies by other groups have shown that synapse strength can be improved temporarily after a short period of paired stimulation between the brain (motor cortex) and the peripheral nerves serving target muscles - in other words, "Fire Together, Wire Together".

The brain's intention to move a muscle can be read by recording surface electrical activity over target muscles (electromyography or EMG). In animal models of SCI, scientists have successfully used target muscle EMG to trigger spinal cord electrical stimulation pulses while the animals perform physical exercises. Using the body's own signals to trigger nerve stimulation is called "closed-loop stimulation". This might be an optimal method to coordinate brain and nerve activity, especially with the clinical advantage of being possible to combine with physical exercise training. However, whether EMG-triggered closed loop stimulation has the same amount of effect when applied non-invasively in humans is still unknown.

This proposed study is a proof-of-principle to demonstrate the potential of non-invasive closed-loop stimulation in humans with incomplete cervical SCI. We will test different combinations of triggered and non-triggered electrical and magnetic stimulation, and record the short-term effects on nerve transmission and skilled function of hand muscles. This pilot study will be a foundation for future studies combining EMG-triggered stimulation with long-term physical exercise training.

DETAILED DESCRIPTION:
In both animal models and humans with spinal cord injury (SCI), synaptic efficacy between corticospinal axons and spinal motor neurons has improved temporarily after a short period of paired stimulation between motor cortex and spinal or peripheral sites. In a demonstration of closed-loop stimulation in SCI rats, target muscle electromyography (EMG) signals were used to trigger spinal cord electrical stimulation while performing physical retraining. Results showed that EMG-triggered stimulation plus physical retraining led to greater motor recovery than non-triggered stimulation or physical training alone. However, these studies used invasive direct spinal cord stimulation in rodent models. Whether this approach can work non-invasively in humans remains unknown.

Twenty participants (10 able bodied and 10 SCI subjects) will be recruited. Each subject will undergo five different 20-minute interventions. Stimulation will be delivered at the motor cortex via transcranial magnetic stimulation (TMS), the median nerve, or both. Stimulation will occur either while the subject is passively at rest or triggered by reaching endogenous EMG threshold during a pinch task. Outcomes will be measured at baseline and every 20 minutes for one hour after the intervention.

The investigators hypothesize that for at least 20 minutes after stimulation, one session of EMG-triggered stimulation will significantly improve motor evoked potential amplitude, increase cortical silent period duration, and decrease time required to complete a pegboard task compared with one session of passively delivered stimulation. The investigators further hypothesize that EMG triggered median nerve stimulation alone will provide equal or greater benefits as EMG triggered TMS or EMG-triggered paired stimulation.

Hypothesis 1: One session of EMG-triggered stimulation will significantly improve motor evoked potential (MEP) amplitude, increase cortical silent period duration of APB, and decrease time required to complete a manual pegboard task compared with one session of passively delivered stimulation or one session of voluntary contraction alone for at least 20 minutes post-stimulation.

Hypothesis 2: EMG-triggered PNS alone will result in equal or greater effects than EMG triggered TMS or TMS+PNS paired stimulation. This would indicate that EMG triggered PNS might be used as a potential intervention to add during physical training, a setting in which TMS is difficult to apply.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Chronic (more than 12 months since injury) motor-incomplete SCI between neurological levels C2-C8
* Score of 3 or more (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction in left or right hand;
* Detectable F-wave responses of the left or right abductor pollicis brevis (APB) to median nerve stimulation;
* Detectable motor evoked potentials in left or right APB;
* Able to perform thumb-middle finger opposition pinch task with detectable APB EMG muscle activity.

Exclusion Criteria:

* Multiple spinal cord lesions;
* History of seizures;
* Ventilator dependence or patent tracheostomy site;
* Use of medications that significantly lower seizure threshold, such as tricyclic antidepressants, amphetamines, neuroleptics, dalfampridine, and bupropion;
* History of stroke, brain tumor, brain abscess, or multiple sclerosis;
* History of moderate or severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
* History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants, or cardiac pacemaker/defibrillator;
* Significant coronary artery or cardiac conduction disease;
* Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures);
* History of bipolar disorder;
* History of suicide attempt;
* Active psychosis;
* Heavy alcohol consumption (greater than equivalent of 5 oz of liquor) within previous 48 hours;
* Open skin lesions over the face, neck, shoulders, or arms;
* Pregnancy
* Unsuitable for study participation as determined by study physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in motor evoked potential (MEP) amplitude of the abductor pollicis brevis (APB) muscle response to single pulses of TMS | Assessed pre, then 0, 20, 40, and 60 minutes post-intervention.
Hand dexterity | Assessed pre, then 0, 20, 40, and 60 minutes post-intervention.
  Timed performance on a grooved pegboard task.

SECONDARY OUTCOMES:
Grip strength | Assessed pre, then 0, 20, 40, and 60 minutes post-intervention.
  Strength will be quantified using hand-held wireless dynamometry.
Change in the duration of the 'cortical silent period' after TMS stimulation during APB contraction | Assessed pre, then 0, 20, 40, and 60 minutes post-intervention.
F-wave responses of the APB muscle | Assessed pre, then 0, 20, 40, and 60 minutes post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y Harel, MD, PhD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.